CLINICAL TRIAL: NCT06561334
Title: The Socioeconomic Impact of Spasmodic Dysphonia Patients and the Role of Botulinum Toxin
Brief Title: Spasmodic Dysphonia Interviews
Status: Active, not recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B01796
Record Dates: First submitted 2024-07-25; First posted 2024-08-20 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Spasmodic Dysphonia; Quality of Life
Keywords: Qualitative study; Interviews; Quality of life; Spasmodic Dysphonia; Botulinum toxin; Laryngology; Voice disorder
MeSH Terms: conditions — Dysphonia; Voice Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spasmodic Dysphonia patients: Adults diagnosed with Spasmodic Dysphonia who have received at least one botulinum toxin injection.
  Interventions: Procedure: Botulinum toxin injections

INTERVENTIONS:
Procedure: Botulinum toxin injections — Botulinum toxin injection to ease spasms of vocal cord

SUMMARY:
Previous research has shown that patients with voice disorders often have a lower quality of life and struggle with employment. Spasmodic Dysphonia (SD) is a voice disorder that causes abrupt and uncontrollable spasms of the voice box, often resulting in the person having lifelong changes in their voice and speech pattern. The current mainstay of treatment is injecting botulinum toxin (BT) injections into the vocal cord to ease the spasms. The same research team conducted a pilot study in April 2021 on patients with SD. The pilot study used questionnaires and short interviews to understand the livelihood of 10 SD patients. It displayed that SD may impact patients' quality of life. The investigators now aim to run an official research project, ethically approved, to explore the following questions further:

1. Does SD impact the socio-economic lives of its patients? If so, how?
2. What role does BT play in the socio-economic livelihood of SD patients?

To answer these questions, the investigators aim to interview 20 patients with Spasmodic Dysphonia.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with Spasmodic Dysphonia who have received at least one botulinum toxin injection.

Exclusion Criteria:

* Below 18 years of age; additional laryngeal condition(s) severely affecting voice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosed Spasmodic Dysphonia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Does Spasmodic Dysphonia impact the socio-economic lives of its patients? If so, how? | Through study completion, which is expected to be a year
  Outcome will be measured through qualitative analysis of participant answers regarding how the target condition, spasmodic dysphonia, affects the social and economic aspects of their livelihood.

SECONDARY OUTCOMES:
What role do botulinum toxin injections play in the socio-economic livelihood of Spasmodic Dysphonia patients? | Through study completion, which is expected to be a year
  Outcome will be measured through qualitative analysis of participant answers regarding how receiving Botulinum toxin injections may improve their livelihood.

CONTACTS AND LOCATIONS:
Overall Officials: Sadie Khwaja, MBChB, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the study content and the interview study design